CLINICAL TRIAL: NCT05073081
Title: Feasibility Testing of a Pre-surgical Rehabilitation (Prehab) Program for Patients With Lumbar Spinal Stenosis: a Pilot Randomized Controlled Trial
Brief Title: Feasibility of Prehab for Lumbar Spinal Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: University of Calgary (Other); University of Alberta (Other)
Responsible Party: Principal Investigator, Luciana Macedo, Assistant Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prehab LSS
Record Dates: First submitted 2021-09-27; First posted 2021-10-11 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Lumbar Spinal Stenosis; Prehabilitation
Keywords: Prehabilitation; Spinal stenosis; Surgery; Exercise therapy
MeSH Terms: conditions — Spinal Stenosis | interventions — lanosterol synthase

STUDY DESIGN:
Intervention Model Description: This is a mixed methods two-armed pilot RCT evaluating an 8-week virtual prehabilitation program for participants undergoing LSS surgery versus usual care. A longitudinal qualitative study will be conducted parallel to the pilot RCT.
Masking Description: Blinding of participants and those delivering the intervention is not possible within rehabilitation trials and blinding of assessors is not possible when participants are not blinded, and outcomes are self-reported. Research coordinators involved in data collection and researchers involved in data analysis, however, will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation (Experimental): The 8-week prehabilitation program will be delivered online using synchronous and asynchronous sessions delivered by either a physiotherapist, chiropractor or kinesiologist. There will be 4 individual exercises sessions delivered synchronously using Zoom or Physitrack in which motivational interviewing and graded activity exercises will be conducted. Participants will also be asked to exercise at least 3 times a week using the asynchronous exercise videos. The exercises will be individualized on participants functional ability and personal goals identified at baseline, with a focus on muscle strengthening, stretching, improving spinal flexibility and stability. There will be a booster session at 6-weeks post-op. Participants will also undergo 5 group educational sessions, which will provide information regarding: goal setting, pain education, self-management, pacing, post-operative expectations, exercise recommendations, and information regarding their upcoming surgery.
  Interventions: Other: Prehab for LSS
- Usual Care (Active Comparator): Participants in the control group will receive usual care as per surgeons' current practice. This generally consists of one session with an anesthesiologist, a nurse and access to our online videos.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Prehab for LSS — The 8-week prehabilitation program will be delivered online by physiotherapists, chiropractors, and kinesiologists through synchronous and asynchronous exercise sessions, along with online educational sessions.
  Arms: Prehabilitation
Other: Usual Care — Participants in the control group will receive usual care as per surgeons' current practice.
  Arms: Usual Care

SUMMARY:
The literature has shown evidence of the effectiveness of prehabilitation programs on post-operative recovery for musculoskeletal conditions; however, evidence for prehabilitation for lumbar spinal stenosis (LSS) is limited. Investigators have found that there is very low to low quality evidence for the effect of prehabilitation interventions for improving outcomes following lumbar spine surgery. Therefore, the purpose of this study will be to determine the feasibility of a prehabilitation program for patients undergoing LSS surgery, and pilot test the protocol to provide the foundation for future design of a larger, multicenter randomized controlled trial.

DETAILED DESCRIPTION:
Background:

Lumbar spinal stenosis (LSS) is the most common degenerative condition among older adults, and the leading reason older adults aged 65 and older undergo surgery. LSS is characterized by degenerative changes that lead to loss of intervertebral disc spaces, joint thickening, and enfolding of the ligaments surrounding the spine. These degenerative changes may cause compression of lumbosacral nerve roots resulting in the narrowing of central and vertebral canals known as neurogenic claudication (NC). The symptoms of NC include cramping, numbness or tingling, and muscle weakness in the lower back, buttocks, or one or both legs, with symptoms often intensifying with standing and walking.

The majority of individuals undergoing surgery for LSS are post-retirement age, have chronic low back pain, without access to private rehabilitation. This population is often severely deconditioned prior to surgery with weakness and atrophy of the muscles in the back, core, and lower limb. These preoperative factors have been shown to be predictors for postoperative LSS outcomes. Studies have shown evidence of the effectiveness of prehabilitation programs on post-operative recovery for other musculoskeletal conditions such as total knee arthroplasty. However, there appears to be a lack of high-quality evidence for the effect of prehabilitation interventions in improving outcomes for LSS surgery.

Research Aims:

The purpose of this study is to determine the feasibility of the program of care on a group of patients with LSS undergoing surgery, and determine the feasibility of the protocol for a randomized controlled trial.

Methods:

This mixed methods study will include a two-armed, pilot RCT evaluating an 8-week virtual prehabilitation program for participants undergoing LSS surgery, with a longitudinal qualitative study conducted parallel to the pilot RCT. The two groups in the RCT study will be: 1) prehabilitation, and 2) usual care.

Recruitment:

There will be 60 participants recruited from participating spine surgeons in 3 Canadian cities - Hamilton, Edmonton, and Calgary. Participants will be included if 1) they are a minimum 20 weeks prior to their date of surgery, 2) older than 55 years of age, 3) are scheduled for first spine surgery , and 4) are English-speaking. Participants will be excluded if 1) they have a known or suspected pathology (e.g., cancer, cauda equina syndrome), 2) are unable to engage in exercise due to other comorbidities or cognitive issues, and 3) if they do not have access to the Internet.

Interventions:

The 8-week prehabilitation program will be delivered online using synchronous and asynchronous sessions delivered by either a physiotherapist, chiropractor or kinesiologist, with a booster session at 6-weeks post-op. There will be 4 individual exercises sessions (week 1, 2, 4 and 8) delivered synchronously using Zoom or Physitrack in which motivational interviewing and graded activity exercises will be conducted. Participants will also be asked to exercise at least 3 times a week using the asynchronous exercise videos. Participants will receive short online educational videos (3-5 minutes). Educational sessions will include information regarding the importance of exercise, pain education, self-management, exercising despite pain, post-operative expectations, and information regarding their upcoming surgery. The educational sessions will also include two online peer-support groups when they can interact with a patient with a history of LSS surgery.

Participants in the control group will receive usual care for LSS surgery, which will consist of one session with an anesthesiologist, a nurse and access to our online educational videos.

Outcomes:

Outcomes will be evaluated at: baseline (~20 weeks before LSS surgery), immediately after the intervention (8-weeks), 3 and 12 months post-operatively. Feasibility outcomes are: 1) recruitment rate; 2) patient adherence to the program and attrition rates; 3) acceptability of program content; and 4); acceptability of study procedures and completion of study questionnaires. Patient reported outcomes will be used to inform feasibility, study burden and sample size calculations. These outcomes include: pain and disability, health-related quality of life, psychological measures, and monitoring variables. Ecological Momentary Assessments using activity monitors will be used to evaluate walking ability and daily pain.

Qualitative Methods A longitudinal qualitative study will be conducted parallel to the pilot RCT. We will use purposive sampling to conduct in-depth semi structured interviews at baseline (~20 weeks before LSS surgery), 8-weeks after the intervention, 3 months, and 12 months post-operatively. For the qualitative study, we will aim to recruit 12-15 participants or until saturation is met. The longitudinal qualitative study will assess the barriers and facilitators that influence engagement in prehabilitation, as well as the changes in pain and health that occur over time and how these are related to the program, personal (e.g., sex and gender, age, comorbid health, pain profile) or contextual factors (psychosocial, environmental, health systems).

Analysis:

All analyses will be conducted using STATA 15. Descriptive statistics will be used to report feasibility outcomes, as well as to identify trends in patient-reported outcomes. Qualitative interviews will be analyzed using interpretive phenomenological analysis (IPA) informed by the Consolidated Criteria for Reporting Qualitative Studies. Inductive thematic analysis will be used to analyze the data and report the study findings.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 20 weeks prior to date of LSS surgery
* Older than 55 years of age
* Scheduled for first spinal surgery
* Can read and understanding English, with no significant visual or hearing impairment that would require additional support

Exclusion Criteria:

* Known or suspected pathology (e.g., cancer, cauda equina syndrome)
* Unable to engage in exercise due to other comorbidities
* No access to the Internet

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Patient Adherence | During the 8-week Intervention
  Measured by patient diary, app-based program
  1. Proceed with study if 80% of participants attended all 4 exercise sessions
  2. Proceed with study if 60% of participants report exercise at last 3x/week.
Recruitment Rate | 20 weeks before LSS surgery
  Proceed with study if 50% of eligible participants consent to participate within 4 months
Content Acceptability | Immediately after the intervention (8-weeks)
  Measured using a survey administered at the end of the 8-week intervention
  1. Proceed with the study if 60% found treatment useful (>7/10 on a Likert scale)
  2. Proceed with the study if 60% found treatment helpful (>7/10 on a Likert scale)
Format Acceptability | Immediately after the intervention (8-weeks)
  Measured using a survey administered at the end of the 8-week intervention
  1. Proceed with the study if 60% found treatment delivery acceptability (>7/10 on a Likert scale)
  2. Proceed with the study if 60% of participants reported being likely to recommend this treatment (>7/10 on a Likert scale)
  3. Proceed with the study if 60% reported being likely to use this treatment again (>7/10 on a Likert scale)
Follow-up | Immediately after the intervention (8-weeks), 3-, and 12-months post-operatively
  1. Proceed with the study if 90% of participants follow-up at the end of the prehab intervention
  2. Proceed with the study if 85% of participants follow-up at 6 months
  3. Proceed with the study if 85% of participants follow-up at 12 months
  4. Proceed with the study if 60% reported being likely to use this treatment again (>7/10 on a Likert scale)
Burden | Immediately after the intervention (8-weeks)
  Proceed with the study if 60% reported being likely to use this treatment again (>7/10 on a Likert scale)

SECONDARY OUTCOMES:
The Oswestry Disability Index | 20 weeks before LSS surgery, immediately after the intervention (8-weeks), 3-, and 12-months post-operatively
  Disease specific questionnaire designed to evaluate pain and function in this patient population, using a numerical rating scale.
Swiss Spinal Stenosis Questionnaire - Balance | 20 weeks before LSS surgery, immediately after the intervention (8-weeks), 3-, and 12-months post-operatively
  Disease specific questionnaire designed to evaluate pain and function in this patient population.
SF-12 | 20 weeks before LSS surgery, immediately after the intervention (8-weeks), 3-, and 12-months post-operatively
  12-Item scale to assess the impact of health on quality of life.
Patient Health Questionnaire-9 | 20 weeks before LSS surgery, immediately after the intervention (8-weeks), 3-, and 12-months post-operatively
  Depression scale to monitor the severity of depression; total score from 0-27 with higher scores representing severe depression.
Pain Catastrophizing Scale | 20 weeks before LSS surgery, immediately after the intervention (8-weeks), 3-, and 12-months post-operatively
  13-item scale to assess the extent of catastrophic thinking due to low back pain. Total score ranging from 0-52, along with three subscale scores assessing rumination, magnification and helplessness.
6-item Chronic Disease Self-Efficacy Scale | 20 weeks before LSS surgery, immediately after the intervention (8-weeks), 3-, and 12-months post-operatively
  6-item scale to evaluate disease related self-efficacy with higher scores indicating higher self-efficacy ranging from 0-10.
Tampa Scale of Kinesiophobia | 20 weeks before LSS surgery, immediately after the intervention (8-weeks), 3-, and 12-months post-operatively
  11-item scale used to evaluate kinesiophobia and associated anxiety. Scores range from 17-68 with higher scores indicating severe kinesiophobia.
Ecological Momentary Assessment | During the 8-week Intervention
  Total weekly minutes of physical activity (PA) will be captured with a wearable tri-axial accelerometer device (Actiwatch Spectrum Pro Startup, Philips, USA) worn for seven consecutive days. Pain and fatigue will be measured using a 10-point scale with higher scores representing worse pain and fatigue, which will be measured 3 times a day for 7 days.
EQ-5D | 20 weeks before LSS surgery, immediately after the intervention (8-weeks), 3-, and 12-months post-operatively
  Measures five dimensions of patient reported health (mobility, self-care, usual activities, pain/discomfort and anxiety/depression).

CONTACTS AND LOCATIONS:
Overall Officials: Luciana G Macedo, PhD, Principal Investigator — McMaster University; Doug Gross, PhD, Principal Investigator — University of Alberta; Lisa Carlesso, PhD, Principal Investigator — McMaster University; Kenneth Thomas, MD, Principal Investigator — University of Calgary
Locations (4):
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - University of Toronto, Toronto, Ontario
  - University of Alberta, Edmonton
  - McMaster University, Hamilton

IPD SHARING:
Plan to Share IPD: Yes
Data may be requested directly to the principal investigator or may be made available upon publication.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available following publication of the results, and kept for at least 5 years to allow for the publication of findings.
Access Criteria: Ethics approval will be required for any secondary analysis of data as per HiREB approval.